CLINICAL TRIAL: NCT01173458
Title: A Multicenter Pilot Study Examining the Role of Circulating Tumor Cells (CTCs) as a Blood-based Tumor Marker in Patients With Small Cell Lung Cancer (SCLC)
Brief Title: Circulating Tumor Cells (CTCs) as a Blood-based Tumor Marker in Patients With Small Cell Lung Cancer (SCLC)
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency); University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 12216
Record Dates: First submitted 2010-07-27; First posted 2010-08-02 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Small Cell Lung Cancer
Keywords: cancer; lung; small cell
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected before treatment begins, at completion of treatment, and every 6 to 8 weeks during follow-up visits.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood Draw: Approximately 1 and one-half teaspoons of blood will be drawn at times specified.
  * one sample prior to treatment initiation
  * one sample after completion of treatment
  * one sample every 6 to 8 weeks during follow up visits
  * one sample at the time of Relapse

SUMMARY:
The purpose of this study is to determine whether or not CTCs can be detected in blood samples taken from patients diagnosed with small cell lung cancer. The purpose is to compare CTC analysis to tumor samples to look for differences.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) is characterized by early dissemination through the blood system with the majority of patients succumbing to their disease in 9-11 months. Despite evaluation of multiple new agents a platinum doublet has remained the standard of care for over 25 years. We believe that the lack of understanding of the biology of SCLC has contributed to our failure to advance treatment and prolong survival. Tumor and blood biomarkers have been shown to be a powerful tool for increasing our understanding of the complex biology of cancer and determining prognosis and response to therapies. Currently, there are no validated biomarkers for response or to follow disease activity in SCLC. Detection of Circulating Tumor Cells (CTCs) is a laboratory technique that became available in the last few decades. Newer, more sensitive technology for the isolation and characterization of CTCs using a rare event imaging system with automated fluorescence microscopy known as CellSearch has demonstrated value in several cancers. CTCs detection by this system is approved as a prognostic biomarker in metastatic breast cancer, and as a tool to monitor disease in metastatic colorectal cancer and castrate resistant prostate cancer.

To date, only one publication has reported on the presence of CTCs in SCLC. These investigators used RT-PCR to amplify CK19 cDNA. CTCs were detected in 27% of patients. In our preliminary study using the CellSearch system we have detected 1 or more CTCs in 11/13 (84%) patient samples in various stages of their disease. Thus CTCs may be a promising biomarker but we need more studies. Thus, our first goal is to determine if CTCs in SCLC can predict response to chemotherapy, predict early relapse or function as a as a prognostic marker.

In addition, we will explore the feasibility of extracting genetic material from CTCs for genomic profile that could immensely help us unravel the complex molecular pathways and gene expression in SCLC, which ultimately will lead to novel drug development. Other investigators have shown that gene expression profiles for CTCs may be used to distinguish normal donor from advanced cancer patients and differentiate among different types of cancers.

In summary, SCLC kills 45,000 Americans each year. The treatment of SCLC has not changed since the introduction of cisplatin and etoposide during 1970s. Research in cancer biology has identified several genetic alterations that could be of therapeutic importance. Novel agents that target these genetic alterations are currently in development. Patient selection will be key in order to determine the activity of these agents. Understanding the biology of this disease is the key to successful interventions and personalizing therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of small cell lung cancer with extensive stage disease and have been untreated.
* Must be willing to give and sign informed consent.
* Must be 18 years of age

Exclusion Criteria:

* Less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be approached during their regularly scheduled Cancer Center appointments.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Subject samples will be used to determine the correlation between CTCs in SCLC patients, detected by CellSearch, with treatment outcomes, including response to chemotherapy, relapse, and survival | average 2 years

SECONDARY OUTCOMES:
Blood samples will be used to examine the genomic profiles of CTCs and compare them to the original tumor specimen. | average 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chao H Huang, MD, FACP, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Centner, Kansas City, Kansas
  - University of Nebraska & Omaha VA, Omaha, Nebraska